CLINICAL TRIAL: NCT01310114
Title: A Phase 2A, Prospective, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety of Intravenous Infusion of Human Placenta-Derived Cells (PDA001) for the Treatment of Adults Following Ischemic Stroke
Brief Title: Study of Human Placenta-derived Cells (PDA001) to Evaluate the Safety and Effectiveness for Patients With Ischemic Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Celularity Incorporated (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCT-PDA001-SK-001
Record Dates: First submitted 2011-02-25; First posted 2011-03-08 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2016-03

CONDITIONS: Stroke, Acute; Middle Cerebral Artery Stroke; Posterior Cerebral Artery Stroke
Keywords: Human Placenta-Derived Cells; Stem cells; Stroke; PDA001; Celgene; cenplacel-L
MeSH Terms: conditions — Stroke; Infarction, Middle Cerebral Artery; Infarction, Posterior Cerebral Artery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): 1 unit PDA001 [approximately 2 x 108 cells] in 240 mL per infusion on Day 1.
  Interventions: Biological: Human Placenta-Derived Cells PDA001- (cenplacel-L)
- Cohort 2A - Experimental (Experimental): 1 unit PDA001 [approximately 2 x 108 cells] or placebo in 240 mL per infusion on Day 1
  Interventions: Biological: Human Placenta-Derived Cells PDA001- (cenplacel-L); Drug: Placebo
- Cohort 2B - Experimental (Experimental): 4 units PDA001 [approximately 8 x 108 cells] or placebo in 240 mL per infusion on Day 1
  Interventions: Biological: Human Placenta-Derived Cells PDA001- (cenplacel-L); Drug: Placebo

INTERVENTIONS:
Biological: Human Placenta-Derived Cells PDA001- (cenplacel-L) — 240 mL of intravenous infusion
Drug: Placebo — Thawed placebo
  Arms: Cohort 2A - Experimental; Cohort 2B - Experimental

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of Human Placenta-Derived Cells (PDA001) at 3 different dose levels versus placebo (vehicle control) administered intravenously in subjects following ischemic stroke. The secondary objective of the study is to assess the effect of PDA001 on improvement in clinical function following ischemic stroke.

ELIGIBILITY:
Inclusion Criteria

1. Males and females 18 years of age to 80 years of age at the time of signing of the informed consent document.
2. Subject or subject's legal representative must understand and voluntarily sign an informed consent document prior to any study-related assessments/procedures being conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. A female of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 48 ± 24 hours prior to treatment with study therapy. In addition, sexually active FCBP must agree to use two of the following adequate forms of contraception methods simultaneously such as: oral, injectable or implantable hormonal contraception; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner for the duration of the study and the follow-up period. Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with FCBP for the duration of the study and the follow-up period.
5. Diagnosis of stroke involving the middle cerebral artery (MCA) territory (cortical and subcortical) or posterior cerebral artery (PCA) (PCA is limited to 3 subjects per cohort) ischemic stroke confirmed by magnetic resonance imaging (MRI)/ computerized tomography (CT). An ischemic stroke is death of an area of brain tissue (cerebral infarction) resulting from an inadequate supply of blood and oxygen to the brain.
6. National Institute of Health Stroke Scale (NIHSS) score of ≥ 6 but < 20 at the time of screening and infusion. Subject should not have shown rapid improvement (≥ 8 point decrease) or deterioration (≥ 4 point increase) in the score from time of initial evaluation to pre-infusion. To the extent possible, the time from initial screening evaluation to reevaluation will be at least 24 hours.
7. Subject must have had a normal neurologic status prior to ischemic episode defined as the absence of focal or global central neurological or psychiatric deficits of sufficient magnitude that it could not reasonably be expected that the subject could recover to the normal range based on the instruments used to assess the subject's response to treatment. The pre-stroke modified Rankin score should be between 0 and 2 inclusive.
8. Treatment with tissue plasminogen activator (tPA) or Food and Drug Administration (FDA)-approved devices used to restore circulation are allowed but treatment must be completed at least 24 hours prior to administration of PDA001.

Exclusion Criteria

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject or subject's legal representative from signing the informed consent form.
2. Pregnant or lactating females.
3. Any condition, including any medical or neuropsychiatric condition, including the presence of laboratory abnormalities, which in the judgment of the investigator places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study including (but not limited to):

   * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT ) > 2.5 x the upper limit of normal at screening.
   * Serum creatinine concentration >1.5 times the upper limit of normal at screening.
   * Bilirubin or alkaline phosphatase level > 2.5 x the upper limit of normal at screening.
   * Glucose < 50 mg/dL or > 250 mg/dL despite adequate antihyperglycemic treatment.
   * Platelet count < 100 x 109 per liter.
   * History of bacteremia or other serious bacterial or fungal infection requiring treatment with IV antibiotics within 84 days (12 weeks) prior to treatment with study therapy other than a treated urinary tract infection.
   * Known infection with human immunodeficiency virus (HIV).
   * Seropositive for hepatitis C or hepatitis B.
   * Known history of seizures.
4. Severe heart failure or evidence of acute myocardial infarction defined of having at least two of the following three features: (1) Chest pain suggestive of cardiac ischemia; (2)Electrocardiogram (ECG) findings of ST elevation of greater than 0.2 mV in 2 contiguous leads, new onset left bundle branch block, ST segment depression, or T-wave inversion; (3) Elevated troponin I. History of prior myocardial infarction within the previous 6 months.
5. Evidence of prior cerebral hemorrhage or ischemic stroke within the last 3 months or recent intracerebral hematomas by head CT or MRI. This exclusion does not include clinically insignificant petechial hemorrhages.
6. Subjects with only lacunar infarcts on MRI or CT. A lacunar infarct is defined as a small (0.2 to 15 mm in diameter) noncortical infarct caused by occlusion of a single penetrating branch of a large cerebral artery.
7. Persistent hypertension with systolic blood pressure (BP) greater than 185 mmHg or diastolic BP greater than 110 mmHg (mean of 3 consecutive arm cuff readings over 20-30 minutes), not controlled by antihypertensive therapy or requiring nitroprusside for control. Efforts should be made to bring systolic blood pressure (BP) to ≤ 160 or diastolic BP ≤ 100 mmHg at the time of IP administration.
8. Clinically significant pulmonary dysfunction, including severe chronic obstructive pulmonary disease (COPD) and history of lung resection.
9. High clinical suspicion of septic embolus.
10. History of pulmonary emboli or deep vein thrombus
11. History of major trauma at time of stroke
12. History of malignancy within 5 years except basal cell or squamous cell carcinoma of the skin or remote history of cancer now considered cured or positive Pap smear with subsequent negative follow up.
13. Known allergy to bovine or porcine products.
14. Known allergy to both gadolinium and iodine based contrast agents for MRI or CT scan preventing the ability to conduct either one of these procedures.
15. Subject has received an investigational agent -an agent or device not approved by FDA for marketed use in any indication-within 90 days (or 5 half-lives, whichever is longer) prior to treatment with study therapy or planned participation in another therapeutic trial prior to the completion of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety (Type, frequency, severity and potential relationship to study drug of adverse events) | Up to 24 months
  A Treatment-emergent AE was any AE that began or worsened in grade after the start of study drug through 30 days after the last dose of study drug or end of study whichever is later. Treatment related toxicity was one considered by the investigator to be possibly, probably or definitely related to study drug. AEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 on the following scale: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = death. A serious adverse event (SAE) is any AE occurring at any dose that: results in death; is fatal or life-threatening; results in persistent or significant disability or incapacity; requires or prolongs in-patient hospitalization; is a congenital anomaly/birth defect in the offspring of a patient; and constitutes an important medical event.
Clinical response defined by a ≥ 1 point decrease from baseline in the Modified Rankin Scale (mRS) at Day 91 post treatment | Baseline to 91 days
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of participants who have suffered a stroke or other causes of neurological disability, and it has become the most widely used clinical outcome measure for stroke clinical trials. The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
Clinical response defined by a ≥ 1 point decrease from baseline in the Modified Rankin Scale (mRS) at Day 181 post treatment | 181 days
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of participants who have suffered a stroke or other causes of neurological disability, and it has become the most widely used clinical outcome measure for stroke clinical trials. The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.

SECONDARY OUTCOMES:
Clinical response defined by a ≥ 1 point decrease from baseline in the Modified Rankin Scale (mRS) at 24 months post treatment | Up to 24 months
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of participants who have suffered a stroke or other causes of neurological disability, and it has become the most widely used clinical outcome measure for stroke clinical trials. The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead
Clinical response defined as a ≥ 4 point decrease from baseline in the National Institute of Health Stroke Scale (NIHSS) | Up to 24 months
  The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.[1] The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
  Score Stroke Severity:
  0 No Stroke Symptoms 1-4 Minor Stroke 5-15 Moderate Stroke 16-20 Moderate to Severe Stroke 21-42 Severe Stroke
Clinical response defined as a clinically significant improvement (at least 20-point increase from baseline) in the Barthel Index (BI) | Up to 24 months
  The Barthel Index (BI) measures the extent to which a person can function independently and has mobility in their activities of daily living (ADL) ie feeding, bathing, groomig, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. The index also indicates the need for assistance in care. Total possible scores range from 0 - 20, with lower scores indicating increased disability. If used to measure improvement after rehabilitation, changes of more than two points in the total score reflect a probable genuine change, and change on one item from fully dependent to independent is also likely to be reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Monica E Luchi, MD, Study Director — Celularity Incorporated
Locations (1):
- Chattanooga Center for Neurologic Research, Chattanooga, Tennessee, United States